CLINICAL TRIAL: NCT05960864
Title: Chinese Spondyloarthritis Inception Cohort
Brief Title: Chinese Spondyloarthritis Inception Cohort (CESPIC)
Acronym: CESPIC
Status: Not yet recruiting | Type: Observational
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Guangxing Chen, Professor, Director, Southwest Hospital, China
Other Study IDs: CESPIC
Record Dates: First submitted 2023-07-06; First posted 2023-07-27 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Ankylosing Spondylitis (AS) / Radiographic Axial SpA (r-axSpA); Non-radiographic Axial Spondyloarthritis (Nr-axSpA); Axial Psoriatic Arthritis (axPsA); Acute Anterior Uveitis (AAU); Crohn Disease (CD); Ulcerative Colitis (UC); Reactive Arthritis (ReA)
MeSH Terms: conditions — Spondylitis, Ankylosing; Non-Radiographic Axial Spondyloarthritis; Uveitis, Anterior; Crohn Disease; Colitis, Ulcerative; Arthritis, Reactive | interventions — Celecoxib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (7):
- Ankylosing spondylitis: Ankylosing spondylitis according to the modified New York criteria or with the clinical diagnosis of AS/r-axSpA fulfilling the ASAS Classification Criteria AND the mNY criteria plus having the indiaction for starting a bDMARD therapy according to the treating rheumatologist
  Interventions: Drug: Celecoxib
- Non-radiographic axial spondyloarthritis: Patients with clinical characteristics of axial SpA but not fulfilling the modified New York criteria for which radiographic sacroiliitis is essential or with the clinical diagnosis of nr-axSpA fulfilling the ASAS Classification Criteria not fulfilling the mNY criteria and the indiaction for starting a bDMARD therapy according to the treating rheumatologist
  Interventions: Drug: Celecoxib
- Juvenile spondyloarthritis: Patients with juvenile spondyloarthritis (juvenile ankylosing spondylitis, juvenile non-AS-spondyloarthritis).
  Interventions: Drug: Celecoxib
- Crohn's disease: Patients with Crohn's disease
  Interventions: Drug: Celecoxib
- Acute anterior uveitis: Patients with acute anterior uveitis
  Interventions: Drug: Celecoxib
- Axial psoriatic arthritis: Patients with the clinical diagnosis of psoriatic arthritis with axial involvement (sacroiliac joints and/or spine) (axPsA)
  Interventions: Drug: Celecoxib
- Reactive arthritis: Patients with reactive arthritis
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Drug: Celecoxib — If we find any behavior that affects the safety of patients in the experiment, we will stop

SUMMARY:
The Chinese Spondyloarthritis Inception cohort (CESPIC) was started 2000 as a prospective, longitudinal, multicentre, nationwide study in China on patients with early SpA including ankylosing spondylitis (AS, also known as radiographic axial spondyloarthritis) and non-radiographic axial SpA. The objectives of CESPIC are to learn about the course of SpA during the very early stage of the disease, to appropriately assess the outcome including radiographic progression of patients after several years of follow-up, to identify outcome predictors, to assess quality of life, function, and costs (direct and indirect costs). CESPIC has been recently expanded to recruit patients with other forms of SpA / conditions associated with SpA: reactive arthritis, acute anterior uveitis, Crohn's disease as well as with psoriasis / axial psoriatic arthritis.

ELIGIBILITY:
Inclusion Criteria:

Crohn's disease. Acute anterior uveitis. Psoriatic arthritis with axial involvement. Reactive arthritis.

Exclusion Criteria:

Infections, Malignancies, Major cardiovascular events, Lower intestinal perforations Other adverse events

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients included in CESPIC are required to have a definite clinical diagnosis of axial SpA / juvenile SpA (currently only adult patients with radiographic axial SpA = ankylosing spondylitis - AS are recruited) or a definite diagnosis of Crohn's disease or a definite diagnosis of acute anterior uveitis or a definite diagnosis of psoriatic arthritis with axial involvement or a definite diagnosis of reactive arthritis.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
BASDAI | baseline
  The Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) disease activity questionnaire contains six questions regarding subjective symptoms
ASDAS | baseline
  The Ankylosing Spondylitis Disease Activity Score (ASDAS) is a new composite index to assess disease activity in Ankylosing Spondylitis (AS)1. It combines five disease activity variables with only partial overlap, resulting in one single score with better truth (validity), enhanced discriminative capacity and improved sensitivity to change as compared to single-item variables
CRP | baseline
  A c-reactive protein test measures the level of c-reactive protein (CRP) in a sample of your blood. CRP is a protein that your liver makes. Normally, you have low levels of c-reactive protein in your blood. Your liver releases more CRP into your bloodstream if you have inflammation in your body. High levels of CRP may mean you have a serious health condition that causes inflammation.
BASMI | baseline
  BASMI was created to help clinicians accurately assess axial status (through five measurements) of individuals suffering from Ankylosing Spondylitis. The measurements are then interpreted to derive a metrology index to define clinically significant changes in spinal mobility.
BASFI | baseline
  The Bath Ankylosing Spondylitis Functional Index is to determine the degree of functional limitation in patients with the inflammatory autoimmune disease Ankylosing Spondylitis (AS).

SECONDARY OUTCOMES:
ASAS20 | baseline
  The ASAS Response Criteria (ASAS 20) is defined as an improvement of at least 20% and an absolute improvement of at least 10 units on a 0-100 scale in at least three of the following domains: Patient global assessment, Pain assessment, Function (BASFI), and Inflammation (last 2 questions of BASDAI).
ASAS40 | baseline
  The ASAS Response Criteria (ASAS 20) is defined as an improvement of at least 40% and an absolute improvement of at least 10 units on a 0-100 scale in at least three of the following domains: Patient global assessment, Pain assessment, Function (BASFI), and Inflammation (last 2 questions of BASDAI).

IPD SHARING:
Plan to Share IPD: Yes
The Chinese Spondyloarthritis Inception cohort (CESPIC) was started 2000 as a prospective, longitudinal, multicentre, nationwide study in China on patients with early SpA including ankylosing spondylitis (AS, also known as radiographic axial spondyloarthritis) and non-radiographic axial SpA. The objectives of CESPIC are to learn about the course of SpA during the very early stage of the disease, to appropriately assess the outcome including radiographic progression of patients after several years of follow-up, to identify outcome predictors, to assess quality of life, function, and costs (direct and indirect costs). CESPIC has been recently expanded to recruit patients with other forms of SpA / conditions associated with SpA: reactive arthritis, acute anterior uveitis, Crohn's disease as well as with psoriasis / axial psoriatic arthritis.
Supporting Information: CSR

REFERENCES:
- [Result] Rudwaleit M, Haibel H, Baraliakos X, Listing J, Marker-Hermann E, Zeidler H, Braun J, Sieper J. The early disease stage in axial spondylarthritis: results from the German Spondyloarthritis Inception Cohort. Arthritis Rheum. 2009 Mar;60(3):717-27. doi: 10.1002/art.24483. PMID 19248087
- [Result] Poddubnyy DA, Rudwaleit M, Listing J, Braun J, Sieper J. Comparison of a high sensitivity and standard C reactive protein measurement in patients with ankylosing spondylitis and non-radiographic axial spondyloarthritis. Ann Rheum Dis. 2010 Jul;69(7):1338-41. doi: 10.1136/ard.2009.120139. Epub 2010 May 24. PMID 20498207
- [Result] Poddubnyy D, Rudwaleit M, Haibel H, Listing J, Marker-Hermann E, Zeidler H, Braun J, Sieper J. Rates and predictors of radiographic sacroiliitis progression over 2 years in patients with axial spondyloarthritis. Ann Rheum Dis. 2011 Aug;70(8):1369-74. doi: 10.1136/ard.2010.145995. Epub 2011 May 27. PMID 21622969
- [Result] Poddubnyy DA, Marker-Hermann E, Kaluza-Schilling W, Zeidler H, Braun J, Listing J, Sieper J, Rudwaleit M. Relation of HLA-B27, tumor necrosis factor-alpha promoter gene polymorphisms, and T cell cytokine production in ankylosing spondylitis -- a comprehensive genotype-phenotype analysis from an observational cohort. J Rheumatol. 2011 Nov;38(11):2436-41. doi: 10.3899/jrheum.110130. Epub 2011 Sep 1. PMID 21885496